CLINICAL TRIAL: NCT03182621
Title: THINK (Translational Health in Nutrition and Kinesiology) Junior Edition
Brief Title: Comprehensive Versus Traditional Lifestyle Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: University of Tennessee (Other)
Responsible Party: Principal Investigator, Arlette Perry, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20120486
Record Dates: First submitted 2017-06-01; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Obesity; Physical Fitness; Cognitive Function 1, Social
Keywords: Physical Fitness; Body Composition; Executive Cognitive Function
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THINK (Experimental): The Translational Health in Nutrition and Kinesiology (THINK) program will have education and fitness sessions lasting two hours, five times a week for a total of 10 weeks. Sessions will include theory, clinical laboratory activities, and physically active games to facilitate a fun environment to enhance physical and health-related fitness, improve nutrition and exercise knowledge and behaviors, and exercise enjoyment and self-confidence.
  Interventions: Behavioral: THINK
- SPARK (Active Comparator): This The Sports, Play, and Active Recreation for Kids (SPARK) group will receive the traditional YMCA SPARK after-school program. They will undergo the same pre and post testing protocol as the intervention group, but will not receive the THINK program.
  Interventions: Behavioral: SPARK

INTERVENTIONS:
Behavioral: THINK — The THINK curriculum was based on the principles of exercise physiology and health behaviors. Sessions included educational components, concentrating on physiology, nutrition, laboratory experiences, and structured physical fitness activities.
  Arms: THINK
Behavioral: SPARK — traditional YMCA program
  Arms: SPARK

SUMMARY:
Despite recommends that school-based interventions use a comprehensive approach for health promotions; most fitness programs exclusively emphasize physical activity. This study compared the comprehensive Translational Health in Nutrition and Kinesiology (THINK) program to a traditional YMCA program (The Sports, Play, and Active Recreation for Kids (SPARK) fitness curriculum) on measures of physical fitness, body composition, and executive cognitive function outcomes among 105 ethnic minority children (9±1.03 years old) following a 10-week intervention period.

DETAILED DESCRIPTION:
Despite recommendations that school-based interventions use a comprehensive approaches for health promotions; most fitness programs exclusively emphasize physical activity. This study compared the comprehensive Translational Health in Nutrition and Kinesiology (THINK) program to a traditional YMCA program (The Sports, Play, and Active Recreation for Kids (SPARK) fitness curriculum) on measures of physical fitness, body composition, and executive cognitive function outcomes among 105 predominantly, ethnic minority children (9±1.03 years old) following a 10week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this study, subjects had to be between the ages of eight and 12, enrolled in a YMCA program, and able to participate in physical activity. Parents were provided with information packets regarding project details, a parental consent form, and a child assent form. Once the subjects assented and parents consented, a health questionnaire regarding child's age, gender, race/ethnicity, health history and SES was completed.

Exclusion Criteria:

* Subjects with metabolic, cardiovascular, neuromuscular and psychological disorders and with medications that would interfere with testing results were excluded from the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in Aerobic Fitness | Baseline and 10 Weeks
  The National Institute of Medicine Toolbox two-minute Walk Endurance Test was used to measure aerobic fitness
Change in Grip Strength | Baseline and 10 Weeks
  Grip strength was measures using a Jamar plus handgrip dynamometer.
Change in Abdominal Strength | Baseline and 10 Weeks
  The one-minute curl-up test was used to measure abdominal strength and endurance.
Change in Lower Body Strength | Baseline and 10 Weeks
  Lower body strength, specifically for the quadriceps muscle group, was assessed with the wall squat test. A vertical jump test utilizing a Vertec. was used to assess lower body power . The vertical jump test data were used to estimate average power (W) according to the Lewis formula Average Power (W) = √4.9 x mass (kg) x √VJ (m) x 9.81.
Change in Percent Body Fat | Baseline and 10 Weeks
  Body composition and body fat was measured using the Inbody-520 multi-frequency bioimpedance analyzer.
Change in BMIz | Baseline and 10 Weeks
  A CDC growth chart statistical resource was used to calculate BMIz using height, weight, age, and gender.
Change in Visceral Abdominal Fat | Baseline and 10 Weeks
  The Saggital Abdominal Height was used as estimate of visceral abdominal fat using a portable anthropometer.
Change in Waist circumference | Baseline and 10 Weeks
  Waist circumference was used to measure central adiposity with a Gulick body tape measure.

CONTACTS AND LOCATIONS:
Overall Officials: Arlette Perry, PhD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: Yes
Only the study investigators and/or sponsor will monitor the plan for data and safety monitoring for this study. Shared data will be done through encrypted files and file management platform OneDrive.